CLINICAL TRIAL: NCT05108649
Title: Study 2: Impact of Nicotine Messaging on Nicotine Beliefs and Tobacco Use Behavior
Brief Title: Impact of Nicotine Messaging on Beliefs and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Strasser (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH); Rutgers University (Other)
Responsible Party: Sponsor-Investigator, Andrew Strasser, Associate Professor, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: UPCC 06021; R01DA051001 (NIH); 849654 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2021-10-14; First posted 2021-11-05 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Smoking Behaviors; Cigarette Smoking
Keywords: Smoking Behavior
MeSH Terms: conditions — Smoking; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: This project will recruit current, daily, non-menthol cigarette smokers to a 35-day, randomized, factorial design protocol. After a 7-day period of smoking own preferred brand cigarettes, participants will be randomized to a 28-day experimental period and will be randomized to one of four conditions: 1) Nicotine Corrective Messaging (NCM) + Reduced nicotine content (RNC) cigarettes, 2) NCM + normal nicotine content (NNC) cigarettes, 3) Delayed Control Messaging + RNC cigarettes, or 4) Delayed Control Messaging + NNC cigarettes.
Who Masked: Participant
Masking Description: Participants are unblinded to the nicotine content of their cigarette, either normal nicotine content (NNC) cigarettes or reduced nicotine content (RNC) cigarettes. However, participants will not be aware of the messaging condition assignment, either Nicotine Corrective Messaging (NCM) or the Delayed Control Messaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nicotine Corrective Messaging (Experimental): After completing a 7-day baseline period, participants will be randomized to a 28-day experimental period and will view nicotine corrective messaging at each in-person session.
  Interventions: Other: Nicotine Messaging
- Delayed Control Messaging (Experimental): After completing a 7-day baseline period, participants will be randomized to a 28-day experimental period and will not view nicotine messaging until the final study session (Delayed Control Messaging).
  Interventions: Other: Nicotine Messaging
- Normal Nicotine Content (NNC) cigarettes (Experimental): After completing a 7-day baseline period of smoking own brand cigarettes, participants will be randomized to a 28-day experimental period and will receive normal nicotine content cigarettes.
  Interventions: Other: Cigarette Condition
- Reduced Nicotine Content (RNC) cigarettes (Experimental): After completing a 7-day baseline period of smoking own brand cigarettes, participants will be randomized to a 28-day experimental period and will receive reduced nicotine content cigarettes.
  Interventions: Other: Cigarette Condition

INTERVENTIONS:
Other: Nicotine Messaging — After completing a 7-day baseline period, participants will be randomized to a 28-day experimental period and will view nicotine corrective messaging at each in-person session or delayed control messaging at the final study session.
  Arms: Delayed Control Messaging; Nicotine Corrective Messaging
Other: Cigarette Condition — After completing a 7-day period of smoking own brand cigarettes, participants will be randomized to a 28-day experimental period and will receive reduced nicotine content (RNC) cigarettes or normal nicotine content (NNC) cigarettes.
  Arms: Normal Nicotine Content (NNC) cigarettes; Reduced Nicotine Content (RNC) cigarettes

SUMMARY:
The purpose of this study is to examine the effect of nicotine messaging and nicotine content of study cigarettes on nicotine beliefs and subsequent use of tobacco and nicotine products.

DETAILED DESCRIPTION:
This project will utilize a randomized, factorial design trial to examine the effects of nicotine messaging on nicotine harm beliefs and smoking behavior. After a 7-day period of smoking own preferred brand cigarettes, participants will begin a 28-day experimental period and will be randomized to one of four conditions: 1) Nicotine Corrective Messaging (NCM) + Reduced nicotine content (RNC) cigarettes, 2) NCM + normal nicotine content (NNC) cigarettes, 3) Delayed Control Messaging + RNC cigarettes, or 4) Delayed Control Messaging + NNC cigarettes. The investigators will aim to recruit and randomize 160 current, daily cigarette smokers (80 male, 80 female) in a 35-day protocol. Participants will be asked to attend 6 in-person sessions at the Center for Interdisciplinary Research on Nicotine Addiction (CIRNA) on Days 0, 7, 14, 21, 28 & 35. Sessions will occur every 6-8 days.

ELIGIBILITY:
Inclusion Criteria:

* Self-report smoking at least 5 non-menthol, filtered cigarettes per day for at least the last 12 months.
* Not currently undergoing smoking cessation treatment or planning to quit over the duration of the study (~6 weeks).
* Plan to live in the area for the duration of the study.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
* Able to communicate fluently in English (i.e., speaking, writing, and reading).

Exclusion Criteria:

* Smoke menthol cigarettes greater than 20% of the time.
* Smoke cigarettes of non-standard circumference (e.g., wides, slim, capri, etc.)
* Use of any nicotine containing products other than cigarettes. Participants reporting isolated use of other nicotine containing products less than 5 times per month are eligible to participate.
* Attempt to quit smoking over the duration of the study period.
* Provide a Carbon Monoxide (CO) reading less than 5 parts per million (ppm) at Session 1 (D0).
* History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse. Attendance at alcoholics anonymous or narcotics anonymous meetings will not be considered medical treatment for the purposes of this protocol.
* Current alcohol consumption that exceeds 25 standard drinks/week.
* Women, including all individuals assigned as "female" at birth, who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period.
* Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the proper completion of the study procedures. Notable impairments will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Color blindness.
* Serious or unstable medical condition. Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Lifetime history of schizophrenia, psychosis, and/or bipolar disorder.
* Current diagnosis of active major depression. Participants who maintain a diagnosis of major depression who have not experienced any major depressive episodes in the past 6 months and are stable on antidepressant medication(s) are eligible to participate.

Additional, general reasons for exclusion include:

* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator and/or Study Physician.
* Any circumstance, medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator and/or Study Physician. Participants may be withdrawn for any of the aforementioned reasons at any point throughout the study.
* Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/or Study Physician. Participants may be withdrawn at any point throughout the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, Ph.D., Principal Investigator — University of Pennsylvania; Andrea Villanti, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Center for Interdisciplinary Research for Nicotine Addiction, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adults who currently smoke cigarettes daily from the Philadelphia, PA region. The last participant completed on June 20, 2024.
Pre-assignment Details: Of 99 participants screened eligible between 3/1/2022 and 6/20/2024, 75% (N = 74) were randomized to one of the four study conditions.
Groups:
- Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will receive normal nicotine content cigarettes, but will not view nicotine messaging until the final study session.
- Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will receive reduced nicotine content cigarettes, but will not view nicotine messaging until the final study session.
- Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will view nicotine corrective messaging at each in-person session and receive normal nicotine content cigarettes.
- Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will view nicotine corrective messaging at each in-person session and receive reduced nicotine content cigarettes.
Period: Overall Study
Arm/Group | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Started | 18 | 19 | 17 | 20
Completed | 16 | 11 | 14 | 12
Not Completed | 2 | 8 | 3 | 8
Not completed — Lost to Follow-up | 0 | 4 | 3 | 6
Not completed — Not Interested | 1 | 1 | 0 | 1
Not completed — Out of area | 0 | 0 | 0 | 1
Not completed — PI decision | 1 | 0 | 0 | 0
Not completed — Significant Non-Compliance | 0 | 1 | 0 | 0
Not completed — Unable to adhere to study protocol | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 18 | 19 | 17 | 20 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.9) | 49.6 (14.1) | 51.2 (12.4) | 49.8 (12.2) | 49.1 (12.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female, Male: Female | 6 | 6 | 4 | 8 | 24
  Sex: Female, Male: Male | 12 | 13 | 12 | 12 | 49
  Sex: Female, Male: Refused | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3 | 6
  Not Hispanic or Latino | 15 | 19 | 16 | 17 | 67
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 4 | 4 | 18
  White | 12 | 12 | 13 | 15 | 52
  More than one race | 1 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Cigarettes per Day [Mean (Standard Deviation); unit: cigarettes per day] | 12.6 (4.6) | 14.7 (6.3) | 13.0 (6.5) | 15.0 (8.0) | 13.9 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Beliefs
Description: Nicotine belief measures will be assessed by participant self-report and comprised of four broad constructs (nicotine beliefs, NRT beliefs, e-cigarette beliefs, and RNC cigarette beliefs). Nicotine beliefs relate specifically to its addictive nature, nicotine as a cause of cancer, and the role of nicotine in the health harms and cancer caused by smoking. The product-specific constructs (i.e., NRT, e-cigarette, RNC cigarette) include items related to the addictiveness of the product and the perceived health risks of the product compared to regular cigarettes. Three items assessing nicotine false beliefs (range 3-11), 6 items assessing nicotine replacement therapy (NRT) false beliefs (range 4-20), 4 items assessing e-cigarette false beliefs (range 2-14), 11 items assessing reduced nicotine content (RNC) cigarettes false beliefs (range 14-45), and two items assessing beliefs about additive-free and organic tobacco products. Higher scale scores indicate a higher number of false beliefs.
Time Frame: Day 35
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
score on a scale
  Nicotine False Beliefs (range 3-11) | 7.5 (2.6) | 8.1 (2.4) | 5.3 (1.9) | 4.8 (2.2)
  NRT False Beliefs (range 4-20) | 10.8 (1.8) | 10.1 (3.1) | 10.3 (2.8) | 8.7 (1.5)
  E-Cigarette False Beliefs (range 2-14) | 9.6 (2.3) | 9.4 (2.5) | 8.3 (2.8) | 8.2 (2.4)
  Reduced Nicotine Content Cigarette False Beliefs (range 14-45) | 31.3 (6.0) | 31.6 (5.0) | 26.6 (7.2) | 24.2 (5.5)
Statistical Analysis 1: Comparison: Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other — We treated the exposure as a four-level categorical variable with control messaging + NNC cigarettes as the control condition; p = 0.0008, ANOVA; ANOVA compared scale scores across the conditions

2. Secondary Outcome: Daily Cigarette Consumption
Description: Daily cigarette consumption will be assessed by participant self-report and verified through collection of spent filters.
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: cigarettes per day
Groups:
- Delayed Control Messaging + Normal Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will receive normal nicotine content cigarettes, but will not view nicotine messaging until the final study session.
- Delayed Control Messaging + Reduced Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will receive reduced nicotine content cigarettes, but will not view nicotine messaging until the final study session.
- Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will view nicotine corrective messaging at each in-person session and receive normal nicotine content cigarettes.
- Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes: After completing a 7-day baseline period, participants will view nicotine corrective messaging at each in-person session and receive reduced nicotine content cigarettes.
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
cigarettes per day | 13.1 (4.6) | 12.5 (6.2) | 13.4 (6.7) | 13.5 (6.7)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.9804, ANOVA

3. Secondary Outcome: Puff Duration
Description: Total puff duration, the sum of all puff durations per cigarette, will be collected using a standardized video scoring procedure. Participants will be video recorded while smoking each lab cigarette in order to collect smoking topography data.
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
Seconds | 18.3 (6.3) | 21.5 (12.0) | 17.3 (7.9) | 18.4 (7.9)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.6579, ANOVA

4. Secondary Outcome: Carbon Monoxide (CO)
Description: Carbon monoxide (CO; measured in parts per million [ppm]) is a measure of toxicant exposure. Two measures assess daily CO exposure (collected at the onset of each session) and CO boost - the change in CO values before and after smoking a cigarette - estimates smoke exposure due to smoking an individual cigarette.
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: Parts per million
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
Parts per million
  Daily CO Exposure | 14.9 (7.0) | 12.4 (6.0) | 15.6 (11.0) | 15.8 (9.9)
  CO Boost | 5.6 (4.0) | 4.3 (2.5) | 5.1 (3.1) | 6.4 (2.2)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.4208, ANOVA

5. Secondary Outcome: Number of Participants With Intention to Use Tobacco/Nicotine Products
Description: Participants will provide subjective ratings for four items assessing intention to use tobacco cigarettes, e-cigarettes, NRT, and RNC cigarettes during the next 12 months. Adapted from PhenX Toolkit- Susceptibility to Tobacco Products, response options Definitely Yes; Probably Yes; Probably Not; Definitely Not. Outcomes reported for participants reporting Definitely Yes or Probably Yes to each item.
Time Frame: Day 35
Measure: Number; unit: participants
Arm/Group | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
participants
  E-Cigarette/Vape | 3 | 1 | 5 | 1
  Nicotine Replacement Product | 4 | 2 | 3 | 5
  Low Nicotine Cigarette | 8 | 2 | 4 | 5
  Cigarette | 16 | 11 | 14 | 11
Statistical Analysis 1: Comparison: Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.245, Chi-squared

6. Secondary Outcome: Tobacco Use
Description: Description Number of days used tobacco in the past 30 days. Days used summed across eight different nicotine/tobacco products (e.g., tobacco cigarettes, e-cigarettes, cigars, NRT, RNC cigarettes).
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
Days | 30.1 (0.9) | 29.2 (4.9) | 28.4 (6.1) | 29.9 (0.3)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.6396, ANOVA

7. Secondary Outcome: Subjective Cigarette Ratings
Description: Participants will provide subjective ratings of the strength and satisfaction for cigarettes smoked at Day 35 using a 100 mm Visual Analogue Scale (VAS). Anchors are item-specific (strength: 0 = "very weak," 100 = "very strong"), with lower scores indicating less favorable ratings.
Time Frame: Day 35
Population: The analytic sample differs from the overall sample due to item non-response.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
units on a scale
  Satisfaction | 61.5 (22.6) | 36.4 (30.6) | 55.1 (27.0) | 36.3 (22.1)
  Strength: number analyzed (Participants) | 16 | 10 | 14 | 12
  Strength | 61.6 (21.2) | 53.2 (28.4) | 61.7 (24.5) | 36.6 (27.3)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.0235, ANOVA

8. Other Pre Specified Outcome: Behavioral Control
Description: One item assessing confidence to resist smoking cigarettes when others are smoking (1=not at all confident to 4=very confident).
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
Score on a Scale | 2.4 (1.2) | 1.7 (0.9) | 2.3 (1.3) | 2.5 (1.1)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.3564, ANOVA

9. Other Pre Specified Outcome: Nicotine Related Norms
Description: Two items: "How would you describe most people's opinion of using nicotine?" and "Thinking about the people who are important to you, how would you describe their opinion on using nicotine?" with five-point Likert scale responses ranging from "very negative" (1) to "very positive" (5). Higher scores indicate positive norms of using nicotine.
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: Score on a Likert Scale
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
Score on a Likert Scale
  People who are important to you | 2.4 (1.0) | 2.3 (1.1) | 2.5 (0.9) | 2.5 (0.8)
  Most People | 2.3 (1.0) | 2.3 (0.8) | 2.5 (1.1) | 2.0 (0.7)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.6057, ANOVA

10. Other Pre Specified Outcome: Attitudes About Nicotine
Description: Three items on nicotine-related attitudes using semantic differentials across five-point Likert scales. 'Using Nicotine is:' Safe (1) - Dangerous (5); Positive (1) - Negative (5); Good (1) - Bad (5).
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Control Messaging + Normal Nicotine Content Cigarettes | Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
Number analyzed (Participants) | 16 | 11 | 14 | 12
score on a scale
  Safe to Dangerous | 4.2 (0.9) | 4.1 (1.3) | 3.6 (1.2) | 3.6 (1.2)
  Positive to Negative | 4.1 (0.9) | 4.3 (0.9) | 4.1 (1.0) | 4.0 (1.0)
  Good to Bad | 4.3 (0.8) | 4.5 (0.8) | 4.2 (0.9) | 3.7 (1.0)
Statistical Analysis 1: Comparison: Delayed Control Messaging + Normal Nicotine Content Cigarettes vs Delayed Control Messaging + Reduced Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes vs Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes; Test type: Other; p = 0.2304, ANOVA

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Overall, there is minimal risk for serious adverse reactions as a consequence of enrolling in this study. AEs will be collected, assessed, and reported as per the study protocol.
Arm/Group | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 8/16 | 4/11 | 4/14 | 10/12
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/11 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 8/16 | 4/11 | 4/14 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes (N=16) | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes (N=11) | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes (N=14) | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes (N=12)
Abscess on right arm (Infections and infestations) | 1 (1) | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Delayed Control Messaging + Normal Nicotine Content Cigarettes (N=16) | Experimental: Delayed Control Messaging + Reduced Nicotine Content Cigarettes (N=11) | Experimental: Nicotine Corrective Messaging + Normal Nicotine Content Cigarettes (N=14) | Experimental: Nicotine Corrective Messaging + Reduced Nicotine Content Cigarettes (N=12)
Sore Throat (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Teeth Extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nausea (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Neck Pain, Shoulder Pain
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Body Aches (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT05108649/Prot_SAP_000.pdf